CLINICAL TRIAL: NCT02325934
Title: Bioequivalence of Crushed Stribild With a Normal Breakfast or With Drip Feed Compared to the Whole Tablet
Acronym: CRUSTRI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: UMCN AKF 14.03
Record Dates: First submitted 2014-10-27; First posted 2014-12-25 (Estimated); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: HIV
Keywords: Stribild; pharmacokinetics; Crushing; Drip feed
MeSH Terms: conditions — Pressure Ulcer | interventions — Elvitegravir, Cobicistat, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Reference (Active Comparator): Stribild Standardized breakfast followed by a single dose of STB (whole tablet).
  Interventions: Drug: Stribild
- Intervention I (Experimental): Stribild, crushed Standardized breakfast followed by a single dose of crushed and suspended STB.
  Interventions: Drug: Stribild, crushed
- Intervention II (Experimental): Stribild, crushed 350 mL of drip feed (type) followed by a single dose of crushed and suspended STB.
  Interventions: Drug: Stribild, crushed

INTERVENTIONS:
Drug: Stribild — Elvitegravir, cobicistat, emtricitabine, tenofovir disoproxil
  Arms: Reference
Drug: Stribild, crushed — Crushed Stribild tablet
  Arms: Intervention I; Intervention II

SUMMARY:
Elvitegravir is an HIV-1 integrase inhibitor which is marketed in a fixed dose combination tablet with cobicistat, tenofovir and emtricitabine (Stribild®, referred to as STB). For patients with swallowing difficulties, administration of whole tablets can be problematic and tablets are cut or crushed to ease administration. In addition if HIV patients develop opportunistic infections, patients can become severely ill and may end up on the intensive care. Patients at the intensive care might not be able to swallow medication. Therefore it is useful to know if it is possible to administer STB through a different route, like a feeding tube. If STB can be crushed or dissolved and given through a catheter it is also useful to know if it can be given with drip feed.

Currently there is no information about crushing STB tablets. "Crushing STB tablets into a liquid medium has not been studied and is not recommended" according to the SPC text. Depending on the biopharmaceutical characteristics of a drug formulation, crushing tablets can lead to altered pharmacokinetics of drugs.

It is important to know whether pharmacokinetics are influenced by crushing of tablets as low concentrations are associated with virologic failure. Therefore higher doses might be needed. In addition, higher Cmax and/or exposure can lead to toxicity. As a result therapeutic drug monitoring is advised, or crushing the drug is a contra-indication based on the available data.

It has been shown that simultaneous oral ingestion of antacids and elvitegravir gives a decrease in Cmax and AUC of elvitegravir. This interaction is not shown for co-ingestion with omeprazole. Which makes it unlikely that this interaction is caused by a pH-lowering effect influencing the absorption of elvitegravir. It is probably a local gastrointestinal complexation phenomenon, similar to what has been observed with other HIV integrase inhibitors. A possible pharmacokinetic interaction between elvitegravir and complexation formers may be expected. Especially considering the active binding sites of elvitegravir which bind magnesium metal ion cofactors. Although there is data that STB can be ingested with a protein rich drink, it is unclear if foods or liquids containing high amounts of magnesium or other cations can cause this same interaction.

Therefore this study will be conducted to investigate whether crushed and suspended STB and crushed and suspended STB with drip feed are bioe-quivalent to taking STB as a whole.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 and not older than 55 years at screening.
* Subject does not smoke more than 10 cigarettes, 2 cigars, or 2 pipes per day for at least 3 months prior to Day 1.
* Subject has a Quetelet Index (Body Mass Index) of 18 to 30 kg/m2, extremes included.
* Subject is able and willing to sign the Informed Consent Form prior to screening evaluations.
* Subject is in good age-appropriate health condition as established by medical history, physical examination, electrocardiography, results of biochemistry, haematology and urinalysis testing within 4 weeks prior to day 1. Results of biochemistry, haematology and urinalysis testing should be within the laboratory's reference ranges (see Appendix A). If laboratory results are not within the reference ranges, the subject is in-cluded on condition that the Investigator judges that the deviations are not clinically relevant. This should be clearly recorded.
* Subject has a normal blood pressure and pulse rate, according to the Investigator's judgement.

Exclusion Criteria:

* Creatinine clearance below 70mL/min.
* Documented history of sensitivity/idiosyncrasy to medicinal products or excipients.
* Positive HIV test.
* Positive hepatitis B or C test.
* Pregnant female (as confirmed by an hCG test performed less than 4 weeks before Day 1 or breast-feeding female. Female subjects of childbearing potential without adequate contraception, e.g. hysterec-tomy, bilateral tubal ligation, (non-hormonal) intrauterine device, total abstinence, double barrier methods, or two years post-menopausal. They must agree to take precautions in order to prevent a pregnancy throughout the entire conduct of the study.
* Therapy with any drug (for two weeks preceding Day 1), except for acetaminophen.
* Relevant history or presence of pulmonary disorders (especially COPD), cardiovascular disorders, neurological disorders (especially seizures and migraine), psychiatric disorders, gastro-intestinal disor-ders, renal and hepatic disorders, hormonal disorders (especially dia-betes mellitus), coagulation disorders.
* Relevant history or current condition that might interfere with drug absorption, distribution, metabolism or excretion.
* History of or current abuse of drugs, alcohol or solvents.
* Inability to understand the nature and extent of the study and the pro-cedures required.
* Participation in a drug study within 60 days prior to Day 1.
* Donation of blood within 60 days prior to Day 1.
* Febrile illness within 3 days before Day 1

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-02; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
AUC | up to 32 hours after administration

SECONDARY OUTCOMES:
adverse events | up to 6 weeks in total
  adverse events will be collected up to 6 weeks in total (entire study)

CONTACTS AND LOCATIONS:
Locations (1):
- CRCN, Radboud University Medical Center, Nijmegen, Netherlands

REFERENCES:
- [Result] Jongbloed-de Hoon M, Colbers A, Velthoven-Graafland K, Duisenberg-van Essenberg M, Kruijssen M, Abbink E, van Crevel R, Burger D. Brief Report: Pharmacokinetics of Crushed Elvitegravir Combination Tablet Given With or Without Enteral Nutrition. J Acquir Immune Defic Syndr. 2017 Apr 15;74(5):571-574. doi: 10.1097/QAI.0000000000001296. PMID 28166190
- See also: paper — https://pubmed.ncbi.nlm.nih.gov/28166190/